CLINICAL TRIAL: NCT06486259
Title: Regional Assessment of the Risk of Lung Injury in Ventilated Patients With Similar Lung Load
Brief Title: Regional Assessment of the Risk of Lung Injury in Ventilated Patients
Acronym: RLY
Status: Recruiting | Type: Observational
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, MD, Hospital El Cruce
Other Study IDs: EL CRUCE HOSPITAL
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: ARDS, Human
Keywords: ARDS; VILI; Mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ventral: Ventral half of the lung
  ..
  Interventions: Other: Controlled mechanical ventilation
- Dorsal: Dorsal half of the lung
  Interventions: Other: Controlled mechanical ventilation

INTERVENTIONS:
Other: Controlled mechanical ventilation — Patients were ventilated under similar tidal volume, respiratory rate, and plateau pressure. PEEP was the adjustment variable to reach a similar plateau pressure

SUMMARY:
Specific characteristics of the lung, such as its functional capacity, heterogeneity, and recruitment potential, can influence the development of ventilator-induced lung injury even under safe ventilation conditions. Objective: To evaluate the risk of ventilator-induced lung injury at the regional level in patients with acute respiratory distress syndrome ventilated with similar tidal volumes and inspiratory pressures.

DETAILED DESCRIPTION:
Mechanical ventilation constitutes a crucial resource serving as a bridge to pulmonary recovery in acute respiratory distress syndrome. However, like any medical intervention, it carries risks of adverse effects, both at the pulmonary and systemic levels. Mechanisms involved in the development of ventilator-induced lung injury include excessive stretching and deformation of lung tissues (stress/strain), cyclic opening and closing of alveoli causing shear stress (atelectrauma injury), and the resulting biological response to tissue damage (biotrauma).

To prevent and/or minimize the risk of ventilator-induced lung injury, monitoring of ventilatory mechanics seeks to understand the effects of the ventilatory cycle on the diseased lung. Factors such as tidal volume, plateau pressure, driving pressure, inspiratory flow, respiratory rate, excessive inspiratory effort, and occasionally positive end-expiratory pressure have been directly associated with the mechanism of damage. From an integrative perspective, the concept of mechanical power seeks to encompass most of these factors within a measurable unit thus expressing the energy repeatedly applied to the respiratory system over a unit of time. Mechanical power provides a more comprehensive view of the burden imposed on the lung and can assist in the identification and management of potential risks associated with mechanical ventilation.

However, mechanical power is not the only factor involved in the development of VILI, as factors such as the duration of mechanical ventilation and the conditions specific to the diseased lung also play a role.ventilator-induced lung injury results from the relationship between the load imposed by the ventilator and the inability of the lung parenchyma to tolerate it. Factors such as reduced lung functional capacity, heterogeneity of aeration loss, and instability of collapsed alveoli, among others, can modulate the lung's tolerance to mechanical injury and influence the development of ventilator-induced lung injury . Finally, different regional lung conditions may give rise to the coexistence of different injury mechanisms in the same lung.

Objective: To evaluate different mechanisms of ventilator-induced lung injury at the regional level in patients with acute respiratory distress syndrome ventilated in the supine position with similar lung load.

ELIGIBILITY:
Inclusion Criteria: ARDS patients

-

Exclusion Criteria:Patients with any of the following criteria were excluded:

* History of emphysema, asthma, pneumothorax, or active bronchopulmonary fistula.
* Severe instability at the time of the study defined by at least one of the following indicators: SaO2 ≤ 90%, shock requiring > 0.5 γ/kg/min of noradrenaline, complex arrhythmia, myocardial ischemia, intracranial hypertension refractory despite first-line measures.
* Esophageal pathology contraindicating esophageal balloon placement (esophageal varices, stenosis, trauma or esophageal surgery, tumor) and/or hematemesis.
* Severe coagulopathy (platelet count <20,000/mm3 or INR >4.
* Inability to undergo computed tomography: morbid obesity (>170 kg) or abdominal circumference >200 cm.
* Patients with do-not-resuscitate orders and pregnant women.
* Participation in another research study in the last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory distress syndrome requiring mechanical ventilatory assistanc
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
comparison of regional lung volume | 1 hour
  comparison of regional lung volume in ml

SECONDARY OUTCOMES:
comparison of regional volume of hyperinflated lung | 1 hour
  comparison of regional volume of hyperinflated lung in ml
comparison of regional lung deformation | 1 hour
  comparison of regional lung deformation in percentage
comparison of the amount of unstable lung | 1 hour
  comparison of the amount of unstable lung in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Pistillo, MD, Principal Investigator — Hospital de Alta Complejidad en Red El Cruce Néstor C. Kirchner
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinokurenko VM. [Dependence of dark adaptation on climatic factors]. Voen Med Zh. 1970 Dec;12:62-3. No abstract available. Russian. PMID 5508674
- [Background] Vallejo-Nagera JA. [New dimensions in the physician-patient relations]. An R Acad Nac Med (Madr). 1970;87(3):247-54. No abstract available. Spanish. PMID 5537108
- [Background] Mascheroni D, Kolobow T, Fumagalli R, Moretti MP, Chen V, Buckhold D. Acute respiratory failure following pharmacologically induced hyperventilation: an experimental animal study. Intensive Care Med. 1988;15(1):8-14. doi: 10.1007/BF00255628. PMID 3230208
- [Background] Dreyfuss D, Saumon G. Ventilator-induced lung injury: lessons from experimental studies. Am J Respir Crit Care Med. 1998 Jan;157(1):294-323. doi: 10.1164/ajrccm.157.1.9604014. No abstract available. PMID 9445314
- [Background] Hotchkiss JR Jr, Blanch L, Murias G, Adams AB, Olson DA, Wangensteen OD, Leo PH, Marini JJ. Effects of decreased respiratory frequency on ventilator-induced lung injury. Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):463-8. doi: 10.1164/ajrccm.161.2.9811008. PMID 10673186
- [Background] Fujita Y, Fujino Y, Uchiyama A, Mashimo T, Nishimura M. High peak inspiratory flow can aggravate ventilator-induced lung injury in rabbits. Med Sci Monit. 2007 Apr;13(4):BR95-100. PMID 17392642